CLINICAL TRIAL: NCT02815371
Title: Laser Acupuncture Before and After Embryo Transfer Improves in Vitro Fertilization Outcomes
Brief Title: Laser Acupuncture Before and After Embryo Transfer Improves IVF Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RMA-00-03
Record Dates: First submitted 2016-05-25; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Embryo Implantation

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (4):
- Needle Acupuncture (Experimental): Sterile, disposable needles were inserted into specific acupoints until Deqi sensation was elicited. The needles were retained for 25 minutes before and after embryo transfer.
  Interventions: Procedure: Needle Acupuncture
- Laser Acupuncture (Experimental): Each point was stimulated with a laser (Luminex Laser Therapy System: Medical Laser Systems, Branford, CT) set at 5 joules/cm2 (J/cm2) in continuous mode for 0.10 seconds. Based on various studies, a minimum of 4 J/cm2 produces an improved circulatory effect.
  Interventions: Procedure: Laser Acupuncture
- Sham Laser Acupuncture (Sham Comparator): However, support staff uninvolved in the design of the trial or analysis of the data disarmed the machine, such that no laser irradiation was emitted. This system created an illusion for both the patient and the acupuncturist, and allowed for a truly double blinded control group.
  Interventions: Procedure: Sham Laser Acupuncture
- No Treatment (No Intervention): This control group was not exposed to any additional physical contact or acupuncture related protocol. They were only exposed to dim light and calming music before and after embryo transfer, mimicking the natural waiting room and procedure room setting for all patients undergoing embryo transfer.

INTERVENTIONS:
Procedure: Needle Acupuncture — See above
  Arms: Needle Acupuncture
Procedure: Laser Acupuncture — See above
  Arms: Laser Acupuncture
Procedure: Sham Laser Acupuncture — See above
  Arms: Sham Laser Acupuncture

SUMMARY:
This study evaluated whether laser acupuncture at the time of embryo transfer (following in vitro fertilization) improves implantation rates. Patients were randomized to one of 4 groups at the time of embryo transfer: 1) laser acupuncture, 2) needle acupuncture, 3) sham laser acupuncture, 4) no treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients seeking pregnancy via in vitro fertilization during the study period

Exclusion Criteria:

* Bleeding disorders (due to the possible use of needles)
* Prior exposure to acupuncture
* Preimplantation genetic screening or diagnosis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 803 (Actual)
Dates: Start 2005-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Implantation rate | Approximately 2 weeks after embryo transfer
  Number of gestational sacs seen on ultrasound per embryo transferred

SECONDARY OUTCOMES:
Clinical pregnancy rate | Approximately 3 weeks after embryo transfer
  Number of pregnancies per embryo transfer procedure
Live birth rate | 40 weeks after intervention
  Number of deliveries of at least on live newborn per embryo transfer procedure

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Reproductive Medicine Associates of Connecticut, Norwalk, Connecticut
  - Reproductive Medicines Associates of New Jersey, Morristown, New Jersey